CLINICAL TRIAL: NCT01028976
Title: Obesity, Inflammation and Oxidative Stress
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Gladys Block, Professor Emerita, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DK062378-05
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: C-reactive Protein; Inflammation; Obesity; Oxidative Stress
Keywords: randomized controlled trial; primary prevention; Vitamin C; Antioxidants; C-reactive protein; inflammation; anti-inflammatory agents; obesity
MeSH Terms: conditions — Inflammation; Obesity | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Two tablets, daily, for 8 weeks
  Interventions: Dietary Supplement: Placebo tablet
- Vitamin C (Experimental): Two tablets, daily, for 8 weeks
  Interventions: Dietary Supplement: Vitamin C (ascorbic acid)

INTERVENTIONS:
Dietary Supplement: Vitamin C (ascorbic acid) — 1000 mg/day (two 500-mg tablets), 8 weeks
  Arms: Vitamin C
Dietary Supplement: Placebo tablet — Placebo tablet (two 500-mg tablets), 8 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether or not Vitamin C (1000 mg/day) can reduce markers of inflammation, especially C-reactive protein (CRP), in obese persons with baseline CRP greater than 1 mg/dl.

DETAILED DESCRIPTION:
The long-term objective of this project is to identify nutritional factors that can reduce the inflammatory component of obesity. Therapies to minimize obesity-related comorbidities are needed, and targeting inflammation may help slow the progression of obesity towards cardiovascular disease and insulin resistance.

Adipose tissue is a source of inflammatory cytokines, and obesity is now viewed as a chronic, low-grade inflammatory state. Inflammation itself is a contributor to the chronic diseases associated with obesity. C-reactive protein (CRP) is a key marker of inflammation, and as a downstream marker it provides functional integration of upstream cytokine activation associated with inflammation. We have previously shown that vitamin C, but not vitamin E, reduces CRP in active and passive smokers and in nonsmokers. The reduction is seen primarily in persons with CRP ≥1.0 mg/L, the CDC threshold for elevated cardiovascular disease risk. We also found that 75% of obese nonsmokers had CRP ≥1.0 mg/L.

The important observation of reduction in elevated CRP by vitamin C now needs to be confirmed in a rigorous study with adequate sample size, to permit justifiable conclusions about the potential usefulness of this agent in reducing inflammation in the obese. We will conduct a placebo-controlled, randomized trial in 552 healthy obese individuals with moderate CRP elevations (CRP ≥1.0 mg/L). Participants will be randomized to either 1000 mg/day vitamin C or placebo for a period of 2 months. We will also characterize the pathways through which this effect takes place by measuring cytokines and oxidative stress.

This project is important because if our previous finding is confirmed in this population, it could offer a low-cost alternative to use of statins to reduce inflammation in persons without other risk factors.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30
* hsCRP ≥ 1 mg/L
* Age 18+
* Member of Kaiser Permanente Health Plan of Northern California

Exclusion Criteria:

* Smoker
* Unwilling to discontinue vitamin supplements for study duration
* Unwilling/unable to use acetaminophen in place of OTC anti-inflammatory medications
* Use of certain medications
* History of certain medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
high-sensitivity C-reactive protein | After 8 weeks of intervention

SECONDARY OUTCOMES:
CRP-related markers of inflammation and oxidative stress, including cytokines and F2-isoprostanes. | After 8 weeks of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Gladys Block, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- Kaiser Permanente of Northern California, Division of Research, Oakland, California, United States

REFERENCES:
- [Background] Block G, Jensen CD, Dalvi TB, Norkus EP, Hudes M, Crawford PB, Holland N, Fung EB, Schumacher L, Harmatz P. Vitamin C treatment reduces elevated C-reactive protein. Free Radic Biol Med. 2009 Jan 1;46(1):70-7. doi: 10.1016/j.freeradbiomed.2008.09.030. Epub 2008 Oct 10. PMID 18952164
- [Background] Block G, Jensen C, Dietrich M, Norkus EP, Hudes M, Packer L. Plasma C-reactive protein concentrations in active and passive smokers: influence of antioxidant supplementation. J Am Coll Nutr. 2004 Apr;23(2):141-7. doi: 10.1080/07315724.2004.10719354. PMID 15047680